CLINICAL TRIAL: NCT04625712
Title: Multicenter Prospective Randomized Study to Choose the Optimal Moment of Colecistectomy After Mild Biliary Pancreatitis
Brief Title: Election of the Optimal Moment of Colecistectomy After Mild Biliary Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/41
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Pancreatitis, Acute
MeSH Terms: conditions — Pancreatitis | interventions — Cholecystectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (experimental arm, surgery intervention) (Experimental): Cholecystectomy within the first week after a mild acute biliary pancreatitis.
  Interventions: Procedure: Cholecystectomy
- Group B (active comparator, surgery intervention) (Active Comparator): Cholecystectomy four weeks later a mild acute biliary pancreatitis.
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Cholecystectomy within the first week after a mild acute biliary pancreatitis

SUMMARY:
Introduction Acute pancreatitis is the third gastrointestinal cause of hospital admission. It is estimated that 35-60% have a biliary origin, and most of them are mild.

After a mild acute biliary pancreatitis (ABP), there is a high risk of recurrence of others biliary events. 15-20% of patients will suffer another pancreatitis, cholangitis, choledocolithiasis, or cholecystitis. Therefore, is necessary a definitive treatment.

Although it is suggested to perform cholecystectomy early, there is still insufficient scientific evidence on this subject. All publications have biases and do not allow establish recommendations. In addition, the usual clinical practice tends to postpone the cholecystectomy, because of doubts about the safety of early intervention and for hospital logistical reasons. On the other hand, is discussing if early cholecystectomy carried out more persistence of residual cholelithiasis, explains for the pathophysiology of the ABP.

Finally, it is important to mention, that in our environment 25% of the patients with an ABP are more than 75 years old. There are not any trial that includes this age group.

Objectives Demonstrate that early cholecystectomy is feasible in all patients, including elderly patients, and decreases the number of readmissions for other biliary events.

Material and Methods It is being done a multicenter prospective randomized trial. After an ABP, patients are randomized in two treatment branches. Group A is cholecystectomy within the first week after the ABP. Group B four weeks later.

There are collect data from demographic information, comorbidities, biliary events before the surgery, residual choledocolithiasis, difficulty of the surgical technique, postoperative complications and patients are follow-up for 6 months.

To obtain a representative sample of the population, we consider it appropriate to include all age groups, including patients older than 75 years.

Expected results With this study we pretend to demonstrate that early cholecystectomy is feasible and safe. It does not increase the number of residual choledocolithiasis, and prevents readmissions for new biliary events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of acute mild biliary pancreatitis according to Altanta 2012 criteria.
* Signed informed consent. Exclusion Criteria
* ASA IV.
* Alcohol abuse or chronic pancreatitis.
* Not having assessed the presence of residual choledocolithiasis (cholangioNMR / intraoperative cholangiography)
* Pregnancy.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients presenting morbidity associated with cholescystectomy | 30 days after surgical intervention
  Number of patients with surgical complications

IPD SHARING:
Plan to Share IPD: No